CLINICAL TRIAL: NCT02921685
Title: A Phase 1 Study of MONALIZUMAB (IPH2201), a Humanized Anti CD94/NKG2A Monoclonal Antibody (Mab) Initiated 2 Months After an HLA Matched Allogenic Stem Cell Transplantation (SCT) Prepared With a Reduced Intensity Conditioning
Brief Title: Study of a Humanized Antibody Initiated 2 Months After an HLA Matched Allogenic Stem Cell Transplantation
Acronym: PIRAT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIRAT-IPC 2015-018
Record Dates: First submitted 2016-09-27; First posted 2016-10-03 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — monalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Monalizumab (Experimental): Monalizumab treatment will be initiated 75 to 100 days after hematopoietic stem cells transplantation. Patients will receive a single dose of monalizumab by intravenous route over 1 hour.
  Interventions: Drug: Monalizumab

INTERVENTIONS:
Drug: Monalizumab — Four dose levels will be tested.
  Other Names: anti CD94/NKG2A; IPH2201

SUMMARY:
This study will determine the Maximal Tolerated Dose if any and the recommended dose for phase 2 of monalizumab, a monoclonal antibody directed against the CD94/NKG2A receptor, after allogenic stem cell transplantation. All patients will receive one single intravenous administration of one of the four doses of monalizumab.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (Allo-HSCT) is a curative option for most of hematological malignancies, though the graft-versus-tumor (GVT) effect mediated by immune cells from the donor. However, the use of Allo-HSCT is limited by its toxicity, notably the graft-versus-host disease (GVHD) that is a major cause of non-relapse mortality (NRM). Conditioning regimens dramatically improved during the last fifteen years, with a decrease of both GVHD and NRM rates. Now, disease recurrence after Allo-HSCT is the first cause of treatment failure and remains a concern for approximately 30% of the patients.

Based on a safety immunologic platform (ATG based reduced toxicity conditioning regimens), it is needed to develop post Allo-HSCT strategies to decrease the incidence of relapse. In this context, the modulation of immune cell activity could play a role to prevent relapse. NK cells have a unique capacity to exert potent GVT effects without inducing GVHD. Moreover, NK cells recovery occurs early after Allo-HSCT and NK cells function are not severely impaired by the use of ciclosporin A, that is given for few months after Allo-HSCT as GVHD prophylaxis. Thus, NK cell modulation appears as a viable option for early immune intervention after Allo-HSCT.

Monalizumab (IPH2201), a monoclonal antibody has a non-depleting and purely blocking activity directed with high affinity and specificity against the CD94/NKG2A receptor expressed by subsets of NK cells, activated αβ CD8+ T cells, γδ-T cells and NK T cells. By suppressing the inhibitory signal transduced by NKG2A, IPH2201 enhances the anti-tumor functions, including cytolytic activity of these immune effector cells.The aim of the study is to determine the safety of IPH2201 after allogenic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting a hematological malignancy (acute myeloid leukemia, acute lymphoblastic leukemia, High risk R-IPSS myelodysplastic syndromes, multiple myeloma, chronic lymphoid leukemia, chronic myeloid leukemia, myeloproliferative neoplasm, Hodgkin lymphoma or Non-Hodgkin lymphoma) treated by allogeneic HSCT according to the following parameters :

   * Donor : HLA matched related or unrelated (10/10) donor
   * Graft : peripheral blood stem cells
   * Conditioning : All types of conditioning reduced toxicity conditioning regimens ATG as in-vivo T-cell depletion
   * GVHD prophylaxis by cyclosporine, still ongoing at full dose at the time of the inclusion
2. Patient being in one of the following post-graft situation at the time of inclusion:

   * Acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) patients: in morphological complete remission (CR) with less than 5% bone marrow blast count.
   * High risk R-IPSS myelodysplastic syndromes patients: with at least marrow CR with less than 5% marrow blast count.
   * Multiple myeloma patients: in at least very good partial response.
   * Chronic Lymphoid Leukemia patients: in CR.
   * Chronic Myeloid Leukemia patients: in hematological CR.
   * Myeloproliferative neoplasm patients: no criteria for disease in acceleration phase.
   * Hodgkin lymphoma or Non-Hodgkin lymphoma patients: in CR.
3. Age ≥ 18 and ≤ 70 years
4. ECOG = 0-1 or Karnofsky index ≥ 70%
5. Clinical laboratory values at screening

   * Calculated creatinine clearance (according to MDRD) > 50 ml/min/1.73 m2
   * Independence of red blood cell transfusion
   * Platelet count > 75 x 109/l
   * ANC > 1 x 109/l
   * Bilirubin < 1.5 ULN
   * ALT and AST < 3 ULN
6. Patients (male or female) who accept and are able to use contraceptive methods recognized as highly effective throughout the study and up to 5 months after the drug administration
7. Signed informed consent of the current clinical study, prior to any protocol-specific procedure
8. Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen

Non inclusion Criteria:

1. Previous history of grade ≥ II acute GVHD (Glucksberg classification)
2. Current active disease or positive serology for HIV before grafting, and/or HCV with detectable viremia and/ or HBV with positive Hbs Antigen.
3. Abnormal cardiac status with any of the following :

   * Ejection fraction (measured by ultrasound or radionuclide imaging) < 50%
   * Unstable angina
   * Myocardial infarction within the last 6 months
   * Presence or persistence of documented congestive heart failure (New York Heart Association functional classification III-IV)
   * Arrhythmia requiring treatment and which is not stabilized by the treatment.
   * QTc ≥ 450 ms (M) or 470 ms (F) (Bazett formula)
4. Previous other allogeneic hematopoietic transplantation or solid organ transplantation
5. Any other serious concurrent uncontrolled medical disorder within 4 weeks prior to IPH2201 administration
6. Use of systemic corticosteroids ongoing or within the last 1 week prior IPH2201 admin-istration
7. Use of any investigational agent within 3 months prior to first dosing (except procedure of conditioning regimen including registered drugs combinations, i.e. Busulfan and Fludarabine or Busulfan and Endoxan)
8. History of another malignancy (except, basal cell carcinoma of the skin, or in situ cervix carcinoma, or any other malignancy in complete remission for more than 3 years since the completion of the treatment). However in the case of leukemia or MDS a previous malignancy accountable for the present disease will not be an exclusion criteria if in complete remission for more than 2 years
9. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
10. Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-05-28 (Estimated); Study Completion 2020-04-28 (Estimated)

PRIMARY OUTCOMES:
Occurence ratio of dose-limiting toxicity (DLT) | 4 weeks
  The occurrence of any of these 3 events will lead to the reporting of a Dose Limiting Toxicity:
  * Any Grade ≥ 3 toxicity according to CTCAE attributable to IPH2201 administration, occurring within 4 weeks of IPH2201 administration and considered as relevant by the investigator
  * Any grade ≥ II acute GVHD requiring a treatment by systemic corticosteroids and occurring within 4 weeks of IPH2201 administration.
  * Any grade ≥ moderate chronic GVHD occurring within 4 weeks of IPH2201 administration.

SECONDARY OUTCOMES:
Incidence of acute GVHD of each grade or chronic GVHD of each degree of severity | from D0 to Week 26 after administration of IPH2201 and at 1 year after transplantation
  Safety will be assessed using Glucksberg's classification for acute Graft versus host disease (GVHD) and NIH classification for chronic GVHD.
Probabilities of non-relapse mortality (NRM) | 1 year after the administration of IPH2201
Cumulative incidence of relapse (CIR) | 1 year after administration of IPH2201.
  Efficacy endpoint
Probability of Disease Free Survival (DFS) | 1 year after the administration of IPH2201
  Efficacy endpoint
Probability of Overall survival (OS) | 1 year after the administration of IPH2201
  Efficacy endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Didier BLAISE, MD, PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhônes, France

REFERENCES:
- [Background] Ruggeri L, Urbani E, Andre P, Mancusi A, Tosti A, Topini F, Blery M, Animobono L, Romagne F, Wagtmann N, Velardi A. Effects of anti-NKG2A antibody administration on leukemia and normal hematopoietic cells. Haematologica. 2016 May;101(5):626-33. doi: 10.3324/haematol.2015.135301. Epub 2015 Dec 31. PMID 26721894
- [Background] Godal R, Bachanova V, Gleason M, McCullar V, Yun GH, Cooley S, Verneris MR, McGlave PB, Miller JS. Natural killer cell killing of acute myelogenous leukemia and acute lymphoblastic leukemia blasts by killer cell immunoglobulin-like receptor-negative natural killer cells after NKG2A and LIR-1 blockade. Biol Blood Marrow Transplant. 2010 May;16(5):612-21. doi: 10.1016/j.bbmt.2010.01.019. Epub 2010 Feb 6. PMID 20139023
- [Background] Rathmann S, Glatzel S, Schonberg K, Uhrberg M, Follo M, Schulz-Huotari C, Kaymer M, Veelken H, Finke J, Fisch P. Expansion of NKG2A-LIR1- natural killer cells in HLA-matched, killer cell immunoglobulin-like receptors/HLA-ligand mismatched patients following hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2010 Apr;16(4):469-81. doi: 10.1016/j.bbmt.2009.12.008. Epub 2010 Jan 4. PMID 20044012
- [Background] Pical-Izard C, Crocchiolo R, Granjeaud S, Kochbati E, Just-Landi S, Chabannon C, Frassati C, Picard C, Blaise D, Olive D, Fauriat C. Reconstitution of natural killer cells in HLA-matched HSCT after reduced-intensity conditioning: impact on clinical outcome. Biol Blood Marrow Transplant. 2015 Mar;21(3):429-39. doi: 10.1016/j.bbmt.2014.11.681. Epub 2015 Jan 9. PMID 25579888
- See also: Official web site of the sponsor — http://www.institutpaolicalmettes.fr